CLINICAL TRIAL: NCT01092507
Title: A Controlled Study of the Immunogenicity and Safety of Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) in Comparison With SA14-14-2 Vaccine in Infants and Toddlers in Thailand
Brief Title: A Study of Japanese Encephalitis Chimeric Virus Vaccine Compared With SA14-14-2 Vaccine in Infants and Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JEC07; UTN: U1111-1112-2269 (Other: WHO)
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-11

CONDITIONS: Encephalitis; Japanese Encephalitis
Keywords: Encephalitis; Japanese Encephalitis; Japanese Encephalitis Vaccines; Infant
MeSH Terms: conditions — Encephalitis; Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JE-CV Group (Experimental): Participants will receive one dose of Japanese encephalitis chimeric virus vaccine (JE-CV)
  Interventions: Biological: Japanese encephalitis chimeric virus vaccine (JE-CV)
- SA14-14-2 vaccine Group (Active Comparator): Participants will receive one dose of Japanese encephalitis live vaccine, SA14-14-2 vaccine. (CD.JEVAX®)
  Interventions: Biological: Japanese encephalitis live vaccine (SA14-14-2 vaccine) (CD.JEVAX®)

INTERVENTIONS:
Biological: Japanese encephalitis chimeric virus vaccine (JE-CV) — 0.5 mL, Subcutaneous
  Arms: JE-CV Group
Biological: Japanese encephalitis live vaccine (SA14-14-2 vaccine) (CD.JEVAX®) — 0.5 mL, Subcutaneous
  Arms: SA14-14-2 vaccine Group

SUMMARY:
The purpose of this study is to compare a single dose of Japanese encephalitis (JE) chimeric virus vaccine (JE-CV) with a single dose of SA14-14-2 live vaccine as primary vaccination in infants and toddlers.

Primary Objective:

* To demonstrate the non-inferiority of the antibody response 28 days after vaccine administration of one dose of JE CV (administered on Day 0) compared to the antibody response after one dose of the SA14-14-2 control vaccine (administered on Day 0).

Secondary Objectives:

* To describe the immune response to JE in both vaccine groups in JE-CV virus and SA14-14-2 virus before and after a single dose of JE CV or a single dose of SA14-14-2 vaccine
* To describe the safety profile in all vaccinated subjects up to 28 days and all serious adverse events (SAEs) up to 6 months after vaccination.
* To describe only related SAEs and all death from 6 month to 12-month follow-up.

DETAILED DESCRIPTION:
All participants will receive one injection of their randomized vaccine on Day 0. Follow-up will continue for 12 months after vaccination.

ELIGIBILITY:
Inclusion Criteria :

* Aged 9 to 18 months on the day of inclusion
* In good general health, without significant medical history
* Provision of informed consent form signed by at least one parent or other legally acceptable representative, and by at least one independent witness if required by local regulations
* Subject and parent/legally acceptable representatives able to attend all scheduled visits and comply with all trial procedures
* Completion of vaccinations according to the national immunization schedule.

Exclusion Criteria :

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing any of the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator
* Receipt of blood or blood-derived products in the past 3 months that might interfere with the assessment of the immune response
* Previous vaccination against flavivirus disease, including Japanese encephalitis (JE)
* Administration of any anti-viral within 2 months preceding first vaccination and up to the 4 weeks following the last trial vaccination at Month 3
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination
* Planned receipt of any vaccine from the inclusion up to the 4 weeks following the last trial vaccination
* Planned receipt of any Japanese encephalitis vaccine during the course of the study
* History of central nervous system disorder or disease, including seizures
* History of flavivirus infection (confirmed either clinically, serologically or microbiologically)
* Febrile illness (temperature ≥ 38°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment.

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Thailand (2):
  - Bangkok
  - Khon Kaen

REFERENCES:
- [Derived] Feroldi E, Pancharoen C, Kosalaraksa P, Chokephaibulkit K, Boaz M, Meric C, Hutagalung Y, Bouckenooghe A. Primary immunization of infants and toddlers in Thailand with Japanese encephalitis chimeric virus vaccine in comparison with SA14-14-2: a randomized study of immunogenicity and safety. Pediatr Infect Dis J. 2014 Jun;33(6):643-9. doi: 10.1097/INF.0000000000000276. PMID 24717964
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 07 March 2010 to 27 April 2011 at 3 clinical centers in Thailand.
Pre-assignment Details: A total of 300 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled; 299 were vaccinated.
Groups:
- Japanese Encephalitis Chimeric Vaccine (JE-CV): Participants received a single dose of Japanese encephalitis chimeric vaccine (JE-CV) on Day 0.
- Japanese Encephalitis Live Vaccine (SA14-14-2): Participants received a single dose of Japanese encephalitis live vaccine (SA14-14-2; CD.JEVAX®) on Day 0.
Period: Overall Study
Arm/Group | Japanese Encephalitis Chimeric Vaccine (JE-CV) | Japanese Encephalitis Live Vaccine (SA14-14-2)
Started | 149 | 150
Completed | 147 | 150
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Japanese Encephalitis Chimeric Vaccine (JE-CV) | Japanese Encephalitis Live Vaccine (SA14-14-2) | Total
Number analyzed (Participants) | 149 | 150 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 149 | 150 | 299
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.1 (2.11) | 13.2 (1.89) | 13.2 (2.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 75 | 144
  Male | 80 | 75 | 155
Region of Enrollment [Number; unit: Participants]
  Thailand | 149 | 150 | 299

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Japanese Encephalitis Seroconversion After Vaccination With One Dose of Either Japanese Encephalitis Chimeric Vaccine (JE-CV) or Japanese Encephalitis Live Vaccine (SA14-14-2) (CD.JEVAX®)
Description: Immunogenicity was assessed by the JE-CV virus and the SA14-14-2 virus 50% plaque reduction neutralization test (PRNT50).
  Japanese Encephalitis seroconversion was defined as a pre-vaccination titer <10 1/dil and post-vaccination titer ≥ 10 1/dil; or a pre-vaccination titer ≥ 10 1/dil and a 4-fold increase from pre- to post-vaccination.
Time Frame: Day 0 through Day 28 after vaccination
Population: Japanese encephalitis antibody titers were assessed in all participants with immunogenicity data and who did not have any protocol violations that might have interfered with primary criteria evaluation (Per-Protocol Population)
Measure: Number; unit: Participants
Arm/Group | Japanese Encephalitis Chimeric Vaccine (JE-CV) | Japanese Encephalitis Live Vaccine (SA14-14-2)
Number analyzed (Participants) | 126 | 128
Participants | 125 | 127

2. Secondary Outcome: Number of Participants With Japanese Encephalitis Seroprotection 28 Days After Vaccination With One Dose of Either Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) or Japanese Encephalitis Live Vaccine (SA14-14-2, CD.JEVAX®)
Description: Immunogenicity was assessed by JE-CV virus 50% plaque reduction neutralization test (PRNT50) or SA14-14-2 virus PRNT50.
  Japanese encephalitis seroprotection defined as participant with antibody titer ≥ 1:10 at baseline (D0) and on Day 28, Month 6, and Month 12.
Time Frame: Day 28 post-vaccination
Population: Japanese encephalitis antibody titers were assessed in all participants with any immunogenicity data who did not have any protocol violations that might have interfered with primary criteria evaluation (Per-Protocol Population)
Measure: Number; unit: Participants
Arm/Group | Japanese Encephalitis Chimeric Vaccine (JE-CV) | Japanese Encephalitis Live Vaccine (SA14-14-2)
Number analyzed (Participants) | 127 | 129
Participants
  Day 0, JE-CV PRNT50 (N = 127, 129) | 0 | 0
  Day 28, JE-CV PRNT50 (N = 125, 128) | 125 | 127
  Day 0, SA14-14-2 PRNT50 (N = 125, 128) | 0 | 0
  Day 28, SA14-14-2 PRNT50 (N = 125, 126) | 122 | 123

3. Secondary Outcome: Number of Participants With Seroconversion After Vaccination With Either Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) or Japanese Encephalitis Live Vaccine (SA14-14-2) (CD.JEVAX®)
Description: Immunogenicity was assessed by JE-CV virus 50% plaque reduction neutralization test (PRNT50) or SA14-14-2 virus PRNT50.
  Seroconversion was defined as a pre-vaccination titer < 10 1/dil and post vaccination titer ≥ 10 1/dil, or a pre-vaccination titer ≥ 10 and a 4-fold increase from pre- to post-vaccination.
Time Frame: Day 28 post-vaccination
Population: Antibody titers were assessed in all participants with any immunogenicity data who did not have any protocol violations that might have interfered with primary criteria evaluation (Per-Protocol Population)
Measure: Number; unit: Participants
Arm/Group | Japanese Encephalitis Chimeric Vaccine (JE-CV) | Japanese Encephalitis Live Vaccine (SA14-14-2)
Number analyzed (Participants) | 127 | 129
Participants
  JE-CV PRNT50 (N = 126, 128) | 125 | 127
  SA14-14-2 PRNT50 (N = 124, 125) | 121 | 122

4. Secondary Outcome: Summary of Geometric Mean Titers of Vaccine Antibodies Before and Following One Dose of Vaccination With Either Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) or Japanese Encephalitis Live Vaccine (SA14-14-2; CD.JEVAX®)
Description: Immunogenicity was assessed by JE-CV virus 50% plaque reduction neutralization test (PRNT50) or SA14-14-2 virus PRNT50.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Japanese Encephalitis Chimeric Vaccine (JE-CV) | Japanese Encephalitis Live Vaccine (SA14-14-2)
Number analyzed (Participants) | 127 | 129
Titers
  Day 0, JE-CV PRNT50 (N = 127, 129) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  Day 28, JE-CV PRNT50 (N = 126, 128) | 491 [378 to 638] | 395 [304 to 514]
  Day 0, SA14-14-2 PRNT50 (N = 125, 128) | 5.00 [5.00 to 5.00] | 5.0 [5.0 to 5.0]
  Day 28, SA14-14-2 PRNT50 (N = 125, 126) | 205 [162 to 259] | 190 [152 to 239]

5. Secondary Outcome: Summary of Participants With Japanese Encephalitis Seroprotection After Vaccination With One Dose of Either Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) or Japanese Encephalitis Live Vaccine (SA14-14-2, CD.JEVAX®)
Description: as for outcome 2
Time Frame: Day 28 up to 12 months post-vaccination
Population: Japanese encephalitis antibody titers were assessed in all vaccinated participants with available immunogenicity data (Full Analysis Set)
Measure: Number; unit: Participants
Arm/Group | Japanese Encephalitis Chimeric Vaccine (JE-CV) | Japanese Encephalitis Live Vaccine (SA14-14-2)
Number analyzed (Participants) | 149 | 150
Participants
  Day 0, JE-CV PRNT50 (N = 149, 150) | 6 | 5
  Day 28, JE-CV PRNT50 (N = 146, 148) | 145 | 147
  Month 6, JE-CV PRNT50 (N = 145, 145) | 137 | 141
  Month 12, JE-CV PRNT50 (N = 143, 146) | 126 | 142
  Day 0, SA14-14-2 PRNT50 (N = 147, 149) | 0 | 0
  Day 28, SA14-14-2 PRNT50 (N = 145, 146) | 141 | 142
  Month 6, SA14-14-2 PRNT50 (N = 145, 145) | 122 | 129
  Month 12, SA14-14-2 PRNT50 (N = 142, 144) | 109 | 126

6. Secondary Outcome: Summary of Geometric Mean Titers of Vaccine Antibodies Before and Following One Dose of Vaccination With Either Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) or Japanese Encephalitis Live Vaccine (SA14-14-2; CD.JEVAX®)
Description: Immunogenicity was assessed by JE-CV virus 50% plaque reduction neutralization test (PRNT50) or SA14-14-2 virus PRNT50.
Time Frame: Day 0 (pre-vaccination) and up to 12 months post-vaccination
Population: Japanese encephalitis antibody titers were assessed in all participants that received a vaccine and with available immunogenicity data (Full Analysis Set)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Japanese Encephalitis Chimeric Vaccine (JE-CV) | Japanese Encephalitis Live Vaccine (SA14-14-2)
Number analyzed (Participants) | 149 | 150
Titers
  Day 0, JE-CV PRNT50 (N = 149, 150) | 5.39 [5.05 to 5.74] | 5.29 [4.98 to 5.61]
  Day 28, JE-CV PRNT50 (N = 146, 148) | 507 [395 to 651] | 370 [291 to 470]
  Month 6, JE-CV PRNT50 (N = 145, 145) | 119 [91.7 to 154] | 103 [85.6 to 124]
  Month 12, JE-CV PRNT50 (N = 143, 146) | 97.6 [74.0 to 129] | 121 [96.7 to 151]
  Day 0, SA14-14-2 PRNT50 (N = 147, 149) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Day 28, SA14-14-2 PRNT50 (N = 145, 146) | 198 [158 to 247] | 171 [138 to 212]
  Month 6, SA14-14-2 PRNT50 (N = 145, 145) | 52.7 [41.2 to 67.4] | 51.4 [41.6 to 63.6]
  Month 12, SA14-14-2 PRNT50 (N = 142, 144) | 46.5 [35.8 to 60.4] | 54.8 [43.9 to 68.4]

7. Secondary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reaction Following Vaccination With One Dose of Either Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) or Japanese Encephalitis Live Vaccine (SA14-14-2 Vaccine) (CD.JEVAX®)
Description: Solicited Injection Site Reactions: Tenderness, Erythema, Swelling. Solicited Systemic Reactions: Fever (Temperature), Vomiting, Crying Abnormal, Drowsiness, Appetite Loss, Irritability.
  Grade 3 Reactions defined as: Tenderness - crying when injected limb was moved, or movement of the injected limb was reduced; Erythema and Swelling - ≥ 5 cm; Fever - temperature > 39.5ºC; Vomiting - ≥ 6 episodes per 24 hours or requiring parenteral hydration; Crying Abnormal - > 3 hours; Drowsiness - Sleeping most of the time or difficult to wake up; Appetite loss - refused ≥ 3 feeds or refused most feeds; and Irritability - inconsolable.
Time Frame: Day 0 through Day 14 post-vaccination
Population: Solicited injection site and systemic reactions were assessed in all participants who received a study vaccination and for whom safety data were available, according to the vaccine actually received (Safety Population).
Measure: Number; unit: Participants
Arm/Group | Japanese Encephalitis Chimeric Vaccine (JE-CV) | Japanese Encephalitis Live Vaccine (SA14-14-2)
Number analyzed (Participants) | 147 | 152
Participants
  Any injection site Tenderness | 44 | 57
  Grade 3 injection site Tenderness | 0 | 1
  Any injection site Erythema | 26 | 35
  Grade 3 injection site Erythema | 0 | 0
  Any injection site Swelling | 9 | 12
  Grade 3 injection site Swelling | 0 | 0
  Any Fever | 24 | 33
  Grade 3 Fever | 0 | 1
  Any Vomiting | 21 | 40
  Grade 3 Vomiting | 1 | 2
  Any Crying Abnormal | 28 | 39
  Grade 3 Crying Abnormal | 1 | 2
  Any Drowsiness | 25 | 38
  Grade 3 Drowsiness | 0 | 0
  Any Appetite Loss | 32 | 54
  Grade 3 Appetite Loss | 0 | 3
  Any Irritability | 41 | 58
  Grade 3 Irritability | 0 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from Day 0 (post-vaccination) through 12 months post-vaccination.
Description: Two participants randomized to receive JE-CV received SA14-14-2 vaccine instead. They were analyzed in the Full Analysis Set according to the group to which they were randomized (JE-CV) and in the Safety Analysis Set according to the vaccine actually received (SA14-14-2 vaccine)
Arm/Group | Japanese Encephalitis Chimeric Vaccine (JE-CV) | Japanese Encephalitis Live Vaccine (SA14-14-2)
Serious Adverse Events (participants affected / at risk) | 14/147 | 18/152
Other Adverse Events (participants affected / at risk) | 66/147 | 88/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Japanese Encephalitis Chimeric Vaccine (JE-CV) (N=147) | Japanese Encephalitis Live Vaccine (SA14-14-2) (N=152)
Oesophageal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Dengue Fever (Infections and infestations) | 1 (1) | 1 (1)
Diarrhoea Infectious (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 6 (6) | 1 (1)
Gastroenteritis Rotavirus (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Infection Enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 2 (2) | 1 (1)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 4 (4)
Balanitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Japanese Encephalitis Chimeric Vaccine (JE-CV) (N=147) | Japanese Encephalitis Live Vaccine (SA14-14-2) (N=152)
Vomiting (Gastrointestinal disorders) | 21/146 (21) | 40 (40)
Crying Abnormal (General disorders) | 28/146 (28) | 39 (39)
Injection Site Erythema (General disorders) | 26/146 (26) | 35 (35)
Injection Site Swelling (General disorders) | 9/146 (9) | 12 (12)
Injection Site Tenderness (General disorders) | 44/146 (44) | 57 (57)
Irritability (General disorders) | 41/146 (41) | 58 (58)
Nasopharyngitis (Infections and infestations) | 14 (14) | 10 (12)
Pharyngitis (Infections and infestations) | 4 (4) | 9 (9)
Upper Respiratory Tract Infection (Infections and infestations) | 11 (12) | 31 (35)
Appetite Loss (Metabolism and nutrition disorders) | 32/146 (32) | 54 (54)
Drowsiness (Nervous system disorders) | 25/146 (25) | 38 (38)
Fever (General disorders) | 24 (24) | 33 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications